CLINICAL TRIAL: NCT02474043
Title: A Community-based, Behavioral Intervention to Improve Screening for Hepatitis C Among High-risk Young Adults in Wisconsin
Acronym: Hep-Net
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: AIDS Resource Center of Wisconsin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2013-1360
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C
Keywords: Injection drug use
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Standard health education and prevention counseling by trained staff
  Interventions: Behavioral: Usual Care
- Hep-Net Intervention (Experimental): Computerized tailored behavioral intervention
  Interventions: Behavioral: Hep-Net Intervention; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Hep-Net Intervention — The Hep-Net Intervention is a web-based questionnaire and tailored feedback system designed to increase readiness to change with respect to several behaviors. The behaviors include (1) reducing or quitting drug use; (2) using sterile equipment every time one injects drugs; (3) undergoing screening for hepatitis C; (4) receiving training to use naloxone to prevent death due to opioid overdose.
  Arms: Hep-Net Intervention
Behavioral: Usual Care — Clients receive health education and risk reduction counseling from a trained prevention specialist.

SUMMARY:
The goal of this study is to evaluate the effectiveness of a brief, computerized behavioral intervention for promoting screening for hepatitis C and reducing risky behavior for people who inject drugs (PWID).

DETAILED DESCRIPTION:
People who inject drugs (PWID) are at high risk for hepatitis C virus (HCV) infection if they share contaminated injection equipment with others. Many are infected but are unaware of it, making it likely they will transmit the virus to others if they share contaminated injecting equipment. Problems related to hepatitis C can be avoided if people know their status by getting tested and referred to treatment.

In this study, the investigators will recruit eligible PWID in several cities in Wisconsin using a social networks strategy, in which clients who receive services at a syringe exchange program are asked to refer peers who also inject drugs to participate in the study. All participants will undergo a baseline computerized risk assessment that elicits information about hepatitis C status, previous testing, transmission risk behaviors, and overdose risk. Participants will then be randomly-assigned to receive either standard risk reduction counseling from a prevention specialist, or computerized tailored risk reduction messages that are specific to their reported risk behaviors, attitudes and beliefs. A follow-up assessment will be completed after 3 months to evaluate changes in behavioral risk and intention to undergo HCV screening. A database will be searched to determine which participants returned for HCV screening within 12 months of enrollment, and of those, which ones tested positive for HCV.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* English-speaking
* Reports injection of illicit drugs in the past month

Exclusion Criteria:

* Unable to provide informed consent due to cognitive impairment
* Unwilling to provide personal locator information and consent to be contacted for follow-up after 3 months.
* Currently known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Screening for hepatitis C infection | 12 months
  Participants will be followed for 12 months to determine whether they undergo repeated screening for hepatitis C

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Westergaard, MD, PhD, Principal Investigator — University of Wisconsin, Madison

REFERENCES:
- [Derived] Hochstatter KR, Hull SJ, Sethi AK, Burns ME, Mundt MP, Westergaard RP. Promoting Safe Injection Practices, Substance Use Reduction, Hepatitis C Testing, and Overdose Prevention Among Syringe Service Program Clients Using a Computer-Tailored Intervention: Pilot Randomized Controlled Trial. J Med Internet Res. 2020 Sep 29;22(9):e19703. doi: 10.2196/19703. PMID 32990630
- [Derived] Westergaard RP, Hull SJ, Merkow A, Stephens LK, Hochstatter KR, Olson-Streed HK, Baker LM, Hess TM. Computerized Tailored Interventions to Enhance Prevention and Screening for Hepatitis C Virus Among People Who Inject Drugs: Protocol for a Randomized Pilot Study. JMIR Res Protoc. 2016 Jan 22;5(1):e15. doi: 10.2196/resprot.4830. PMID 26800903